CLINICAL TRIAL: NCT05744583
Title: Finnish Prehospital Whole Blood Study
Acronym: FinnPHWB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Red Cross Blood Service (Other)
Collaborators: Helsinki University Central Hospital (Other); Tampere University Hospital (Other); Päijät Häme Central Hospital (Other)
Responsible Party: Principal Investigator, Jouni Lauronen, Principal Investigator, Finnish Red Cross Blood Service
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FinnPHWB
Record Dates: First submitted 2022-12-23; First posted 2023-02-27 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hemorrhage
Keywords: Transfusion; Prehospital emergency care
MeSH Terms: conditions — Hemorrhage | interventions — Exchange Transfusion, Whole Blood

STUDY DESIGN:
Intervention Model Description: Non-randomized, open label design. 3 centers use whole blood while others use packed red cells as pre-hospital transfusion therapy. Only study related intervention is additional blood samples from sub-group of patients for in vivo coagulation studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Packed red blood cell (Active Comparator): control
  Interventions: Other: Packed red cell transfusion
- Low titer whole blood (Experimental): case
  Interventions: Other: Whole blood transfusion

INTERVENTIONS:
Other: Packed red cell transfusion — Type O RhD negative packed red cell transfusion during prehospital emergency care
  Arms: Packed red blood cell
Other: Whole blood transfusion — Type O RhD positive, low titer whole blood transfusion during prehospital emergency care
  Arms: Low titer whole blood

SUMMARY:
Up-to-date evidence suggests that blood transfusion initiated as early as possible reduces the likelihood of death from hemorrhagic shock, and the sooner replacement therapy with blood products is initiated, the greater the effect on mortality. Typically, the patient is transfused with one to two units of O RhD (Rh blood group D antigen) negative packed red blood cells (PRBC). Hemostasis accelerating medicines (dry plasma, tranexamic acid, calcium, fibrinogen) as well as crystalloids are also often given.

Finnish Red Cross Blood Service is validating cold stored, 0 RhD positive, male donor, leucoreduced, platelet sparing, low blood group ABO antibody titer whole blood product (LTOWB). For this prospective, open, non-randomized clinical study LTOWB will be used in three prehospital emergency medical services that currently use most of prehospital blood products in Finland, while other participating prehospital emergency medical service bases provide controls. Blood transfusions will be given for clinical indication only.

The primary goal is to introduce LTOWB and to analyze its feasibility in Finnish prehospital emergency medical service. Study also aims to prove safety of LTOWB, and to analyze coagulation properties of LTOWB compared to currently prehospitally used PRBC transfusions.

DETAILED DESCRIPTION:
Up-to-date evidence suggests that blood transfusion initiated as early as possible reduces the likelihood of death from hemorrhagic shock, and the sooner replacement therapy with blood products is initiated, the greater the effect on mortality. Since the mid-2010s, prehospital emergency medical services in Finland have used blood transfusions. Typically, the patient is transfused with one to two units of O RhD (Rh blood group D antigen) negative packed red blood cells (PRBC). Hemostasis accelerating medicines (dry plasma, tranexamic acid, calcium, fibrinogen) as well as crystalloids are also often given during pre-hospital emergency treatment. Platelets are not used prehospitally in Finland due to logistic reasons.

The international trend has been the re-emergence of whole blood as the primary replacement product for acute bleeding. Finnish Red Cross Blood Service is validating cold stored, 0 RhD positive, male donor, leucoreduced, platelet sparing, low blood group ABO antibody titer whole blood product (LTOWB). For this prospective, open, non-randomized clinical study LTOWB will be used in three prehospital emergency medical services that currently use most of prehospital blood products in Finland (HUS area, Pirkanmaa area and Päijät-Häme area). Other participating prehospital emergency medical service bases provide controls. Blood transfusions will be given for clinical indication only.

The primary goal is to introduce LTOWB and to analyze its feasibility in Finnish prehospital emergency medical service. Study also aims to prove safety of LTOWB, and to analyze coagulation properties of LTOWB and its effects on endothelial injury and inflammation compared to currently prehospitally used PRBC transfusions. The primary endpoint of the clinical study is the number of patients having severe coagulopathy (measured as INR of = 1.5) at hospital arrival. The secondary outcomes in order of precedence are: Number of patients having coagulopathy at hospital arrival (INR >1.2), time at the scene of transfusion capable unit , need for massive transfusion protocol at hospital, discharge from primary hospital, discharge from intensive care unit, number of patients with acute lung injury according to Berlin definition, in-hospital mortality, 24 hour mortality, any serious adverse effect within 30 days, any adverse effect excluding anti-D formation of D-negative patients within 30 days.

Study begins at first quarter of 2022 and recruiting for clinical part of the study continues three years. All adult (=18 years of age) patients who receive prehospital LTOWB or PRBC transfusion during study period in contributing prehospital emergency medical services will be asked to participate using delayed informed consent procedure from patient, or their next of kin if patient is unable due to his/her condition. Consent will not be asked from next of kin and no blood samples for study will be collected, if patient dies before any contact.

In addition to clinical data, a survey that analyses the emergency care team-members' experiences of transfusion events at prehospital setting will be conducted, and prehospital time logs will be compared between the LTOWB and control groups. In addition, separate blood samples will be collected for coagulation, endothelial injury and inflammatory response analyses from subsample of the patients.

ELIGIBILITY:
Inclusion Criteria:

-All adult patients that have been given a blood transfusion during prehospital emergency care

Exclusion Criteria:

- Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Severe coagulopathy | within 30 minutes upon arrival to the hospital
  Number of patients having severe coagulopathy (measured as INR of = 1.5)

SECONDARY OUTCOMES:
Coagulopathy | within 30 minutes upon arrival to the hospital
  Number of patients having coagulopathy (INR >1.2)
Time spend at the scene | 1-500 minutes
  Time (min) from arrival of transfusion capable unit at the scene to depart of the patient to the hospital.
Number of patients needing massive transfusion protocol | During first 24 hours after arrival to the hospital
  Need for massive transfusion protocol at hospital
Time treated at the hospital | From day 0 (arrival to the hospital) to the date of discharge from the hospital or date of death from any cause, whichever came first, assessed up to 36 months.
  Time (days) patient is treated at the hospital capable of providing curative treatment to the patients medical condition. Data gathered from patient records (admission to ICU and discharge from ICU date)
Time treated at the intensive care unit | From day 0 (arrival to ICU) to the date of discharge/removal to the ward or date of death, whichever came first, assessed up to 36 months.
  Time (days) patient is treated at the intensive care unit during first ICU episode. Data gathered from patient records (admission to ICU and discharge from ICU date)
Number of patients with acute lung injury | From day 0 (arrival to the hospital) to the date of discharge from the hospital or date of death, whichever came first, assessed up to 36 months
  Number of patients with acute lung injury according to Berlin definition
In-hospital mortality | From day 0 (arrival to the hospital) to the date of discharge from the hospital or or date of death, whichever came first, assessed up to 36 months
  Mortality during initial hospitalization period
24 hour mortality | 24 hours from the event
  Any mortality during first 24 hours from event
Serious adverse effects | 30 days from the event
  Any serious adverse effect within 30 days
Adverse effects | 30 days from the event
  Any adverse effect excluding anti-D formation of D-negative patients within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jouni Lauronen, MD, PhD, Principal Investigator — Finnish Red Cross Blood Service
Locations (1):
- PH00, Lahti, Finland